CLINICAL TRIAL: NCT05044208
Title: Echocardiographic Predictors of Atrial Fibrillation in Patients With ESUS or TIA - Detected With 7-day ECG Monitor
Brief Title: Echocardiographic Predictors of Atrial Fibrillation
Acronym: EPAF-7
Status: Recruiting | Type: Observational
Sponsor: Karl Landsteiner University of Health Sciences (Other)
Collaborators: NÖ Landesgesundheitsagentur, legal entity of University Hospitals in Lower Austria (Unknown); Department of Internal Medicine, University Hospital Tulln, Alter Ziegelweg 10, 3430, Tulln, Austria (Unknown); Department of Neurology, University Hospital Tulln, Alter Ziegelweg 10, 3430, Tulln, Austria (Unknown)
Responsible Party: Principal Investigator, Erol Erdik, Principle Investigator, MD, Karl Landsteiner University of Health Sciences
Other Study IDs: 1018/2020
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation; Stroke, Ischemic; Embolic Stroke of Undetermined Source; TIA, Brain
Keywords: Echocardiography; Total Atrial Conduction Time; Left Atrial Strain; Left Atrial Volume
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke; Ischemic Attack, Transient | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No atrial fibrillation detected: In this cohort, AF is not detected in 7-day ECG monitoring or 2-years follow-up period
  Interventions: Diagnostic Test: ECG monitoring
- Atrial fibrillation detected: In this cohort, AF is detected in 7-day ECG monitoring or 2-years follow-up period
  Interventions: Diagnostic Test: ECG monitoring

INTERVENTIONS:
Diagnostic Test: ECG monitoring — After clinical routine diagnostics an additional ambulatory ECG monitoring for 7 days is established

SUMMARY:
This prospective study aims to identify the diagnostic accuracy of echocardiographic predictors of atrial fibrillation in patients with ESUS (embolic stroke of undetermined source) or TIA (transient ischemic attack).

DETAILED DESCRIPTION:
Cardiac thromboembolism attributed to atrial fibrillation (AF), the most frequent cardiac arrhythmia, is responsible for up to one-third of ischemic strokes.

Several factors have been proposed to predict AF, as findings in 12-lead ECG (electrocardiogram) or Holter ECG, epidemiological or echocardiographic parameters.

The main purpose of this research project is to test the diagnostic accuracy of the atrial electromechanical conduction time, measured as septal total atrial conduction time "sPA-TDI", an echocardiographic parameter, and the LaHAsPa-Score, which is based on patient characteristics and echocardiographic measurements for the detection of AF in patients diagnosed with ESUS or TIA, utilizing a 7-day ambulatory ECG monitor and incidental detection of AF during a two-year follow-up period, including detection via implantable cardiac monitor or pacemaker, if applicable.

Other echocardiographic measurements including left atrial volume index (area-length method), atrial electromechanical delay, left atrial myocardial strain together with laboratory, 12-channel ECG, Holter ECG findings, and established risk scores will be compared to the main parameters of interest.

The investigators expect that the results will help with better risk stratification and targeted monitoring periods for atrial fibrillation in patients with ESUS or TIA.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years, written informed consent to participate in the study Clinical diagnosis of ischemic stroke or transient ischemic attack + brain imaging to rule out hemorrhagic stroke.

1. Stroke: ESUS, defined as all of the following:

   * Stroke detected by CT (computertomography) or MRI (magnetic resonance imaging) that is not lacunar. (Lacunar is defined as a subcortical (this includes pons and midbrain) infarct in the distribution of the small, penetrating cerebral arteries whose largest dimension is ≤1.5 cm on CT or ≤2.0 cm on MRI diffusion images/<1.5 cm on T2 weighted MR images. The following are not considered lacunes: multiple simultaneous small deep infarcts, lateral medullary infarcts, and cerebellar infarcts.)
   * Absence of extracranial or intracranial atherosclerosis causing ≥50 percent luminal stenosis of the artery supplying the area of ischemia. Patients must undergo vascular imaging of the extracranial and intracranial vessels using either catheter angiography, CT angiogram (CTA), MR angiogram (MRA), or ultrasound, as considered appropriate by the treating physician and local principal investigator.
   * No major-risk cardioembolic source of embolism, including intracardiac thrombus, mechanical prosthetic cardiac valve, atrial myxoma or other cardiac tumors, mitral stenosis, myocardial infarction within the last 4 weeks, left ventricular ejection fraction <30 percent, valvular vegetations, or infective endocarditis).
   * No other specific cause of stroke identified, such as arteritis, dissection, migraine, vasospasm, drug abuse, or hypercoagulability. Special testing, such as toxicological screens, serological testing for syphilis, and tests for hypercoagulability, will be performed at the discretion of the treating physician and local principal investigator, if needed.
2. TIA: Patients fulfilling all above criteria and diagnostic work-up, except the detection of ischemic lesions by CT or MRI is optional and clinical symptoms last < 1 hours.

All patients must undergo electrocardiogram, transthoracic or transesophageal echocardiography (TTE or TEE) and at least 24 hours of cardiac rhythm monitoring (Holter monitor or telemetry or equivalent).

Patent foramen ovale is not an exclusion criterion. Planned or existing implantation of an implantable cardiac monitor or cardiac pacemaker is not an exclusion criterion.

Exclusion Criteria:

* History of AF, AF on 12-lead ECG, or any AF of any duration during heart-rhythm monitoring prior to inclusion into the study
* Technical problems or bad quality of the echocardiogram making it impossible to measure the main parameters for calculating the LaHAsPa-Score (sPA-TDI, LAVI)
* Wearing time < 1 week (combined recording time < 168 hours) due to patient withdrawing from study, patch dissolving or technical defects
* Life expectancy < 1 month
* Patients under custody or mentally not being able to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are hospitalized with ischemic stroke or TIA at the department of neurology, meet the eligibility criteria and are willing to participate with informed consent
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Detection of former unrecognized atrial fibrillation | 7 days (168 hours of ECG recording)
  AF will be defined as an episode of irregular heart rhythm, without detectable P waves, lasting more than 30 seconds

SECONDARY OUTCOMES:
Detection of atrial fibrillation after 7 days in the follow-up period | 24 months
  participants wearing the device for more than a week or diagnosed with AF after home monitoring period by local physicians or via ICM (implantable cardiac monitor) or pacemaker
Recurrent ischemic stroke | 24 months
  occurence of ischemic stroke during the follow-up period
Participants on oral anticoagulation | 24 months
  participants who have been prescribed oral anticoagulants by their treating physician (for any reason)
Cardiovascular (CV) death | 24 months
  AMI (acute myocardial infarction), sudden cardiac death, death due to heart failure (HF), death due to stroke, death due to CV procedures, death due to CV hemorrhage and other CV causes

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Frank, Professor, Study Director — Head of Internal Medicine Department, University Hospital Tulln
Locations (1):
- University Hospital Tulln, Tulln, Austria

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification
Supporting Information: Study Protocol, ICF, CSR
Time Frame: immediately following publication, no end date
Access Criteria: Proposals should be directed to erol.erdik@tulln.lknoe.at, data access will be granted via a third party website. Anyone who wishes to access the de-identified data for research purposes is eligible.